CLINICAL TRIAL: NCT00000216
Title: Buprenorphine Maintenance for Cocaine Abusing Opioid Addicts
Brief Title: Buprenorphine Maintenance for Cocaine Abusing Opioid Addicts - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Treatment
Other Study IDs: NIDA-06266-1; R01DA006266 (NIH); R01-06266-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Cocaine-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders
Keywords: Opioid-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders; Opioid-Related Disorders; Substance-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to compare the clinical efficacy of maintenance on low and high doses of buprenorphine with methadone for cocaine abusing opiate addicts.

ELIGIBILITY:
Please contact site for information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Depression
Withdrawal symptoms
Opioid and cocaine use
Social and psychological functioning
AIDS risk behavior

CONTACTS AND LOCATIONS:
Overall Officials: Richard Schottenfeld, M.D., Principal Investigator — Yale University
Locations (1):
- APT Residential Services Division, New Haven, Connecticut, United States

REFERENCES:
- [Background] Schottenfeld RS, Pakes JR, Oliveto A, Ziedonis D, Kosten TR. Buprenorphine vs methadone maintenance treatment for concurrent opioid dependence and cocaine abuse. Arch Gen Psychiatry. 1997 Aug;54(8):713-20. doi: 10.1001/archpsyc.1997.01830200041006. PMID 9283506